CLINICAL TRIAL: NCT05908617
Title: Heart Failure Patient Education Using Video and Paper Discharge Instructions
Brief Title: Impact of Video Discharge Instructions on Heart Failure Patient's Knowledge
Acronym: VID-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per PI this QI/QA resident project was not initiated. Record should be deleted.
Sponsor: Yasmeen Golzar (Other Government)
Responsible Party: Sponsor-Investigator, Yasmeen Golzar, Principal Investigator, Cook County Health
Organization: Cook County Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-538-Stroger
Record Dates: First submitted 2018-01-12; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: Patient knowledge; Heart Failure; Self Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper Discharge Instruction (No Intervention): Patient will be given paper discharge instructions
- Video Discharge Instructions (Experimental): Patient will be given Video discharge instructions
  Interventions: Other: Video Discharge

INTERVENTIONS:
Other: Video Discharge — Patient will watch a video discharge instructions in addition to the standard paper instructions. They will also take the pre and post test as the control group
  Arms: Video Discharge Instructions

SUMMARY:
With improve care of patients with heart failure, many patients are living longer. Care for these patients is now not only focused on mortality but also on the quality of life. Patient knowledge about heart failure and their overall compliance with the necessary lifestyle changes will lead to an improved quality of life. Discovering alternative ways to improve patient knowledge is key to long term survival. This studies objective is to assess the overall impact of video discharge instructions as compared to paper discharge instructions on Heart Failure Knowledge among an under-served patient population.

DETAILED DESCRIPTION:
In this study, we will randomized patients admitted to the hospital with heart failure exacerbation to receive either paper or video discharge instructions within a day prior to discharge. The video and paper instructions will have the same content. The patients will take a pre-test and post-test and the change in scores among the patients who received the video and paper discharge instructions will be compared. Other points of interest include participant satisfactions with discharge instruction, followup at post hospital appointment and 30-day readmission.

Data to be collected includes:

1. Medial history of the patient
2. Educational background
3. Social Status
4. Patients Health Measurement: Self Efficacy for managing medications and Treatment Management, Informational Support

ELIGIBILITY:
Inclusion Criteria:

* hospital admission with a diagnosis of Heart Failure (HF)- Heart failure with reduced ejection fraction or heart failure with preserved Ejection fraction
* planned discharge from hospital to home setting
* able to read and write English
* Acceptable to answer Questionnaire and to receive a call at the end of the study

Exclusion Criteria:

* Planned discharge to long term acute care
* Patients with unstable housing
* imprisoned patients
* patients who are pregnant
* illiteracy (defined as inability to write or read) and non-native speakers of English
* impaired cognition
* impaired vision
* Patients with End Stage Renal Disease(ESRD)
* Cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Heart Failure Knowledge Score | 1hr
  Participants knowledge about heart failure will be assessed using the validated Atlanta Heart Failure Knowledge Test(AHFKT- V3). This is a test which includes 30 questions with a minimum score of 0 and a maximum score of 30. Each Participant will take the test and will subsequently be given either paper discharge instructions or both video and paper discharge instructions. After reading and/or watching the discharge instructions, each participant will take the same test once again. The difference in the pre and post intervention scores will be calculated and the investigators will assess if there is a significant difference in the mean change in score the control(Paper) vs. Intervention groups(Video).

SECONDARY OUTCOMES:
Participant Satisfaction with discharge Instructions | 1 day
  Participant overall satisfaction with their discharge instructions will be assess using a 5 point likert scale which ranges from not at all helpful to extremely helpful
Post hospital followup rates | 30 days
  Upon discharge from the hospital, Each participant is given a post hospital appointment within 14 days of the discharge date. We will assess the percentage of participates in both groups who come to post hospital appointments.
Heart Failure Readmission rates | 30days
  Investigators will assess the percentage of participants in both groups who will be readmitted to the hospital within 30days after being discharged from the index visit.

CONTACTS AND LOCATIONS:
Locations (1):
- John H Stroger Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided